CLINICAL TRIAL: NCT01877850
Title: Non Pharmacological Randomized Clinical Trial Designed to Evaluate the Difference of the Duration of Weaning Process From the Ventilator Between Protocol-driven Weaned Patients and Clinical-driven Weaned Patients.
Brief Title: Utility of a Weaning Protocol in ICU
Acronym: WEAN
Status: Completed | Type: Observational
Sponsor: ELENA PELI,MD (Other)
Responsible Party: Sponsor-Investigator, ELENA PELI,MD, dirigente medico, Università degli Studi di Brescia
Organization: Università degli Studi di Brescia (Other)
Other Study IDs: NPn1351
Record Dates: First submitted 2013-06-01; First posted 2013-06-14 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Weaning Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- case: patients with BPAW-M more than 15 or between 10 and 15, but with Tobin <100 will be weaned with the weaning protocol by nurses
  Interventions: Procedure: weaning protocol
- control: patients with any BWAP-M will be weaned by clinical judgment of physicians

INTERVENTIONS:
Procedure: weaning protocol — Reduction of pressure support ventilation (PSV) by 2cmH2O at a time to a maximum of 4cmH2O per day.
  When a patient was able to tolerate PSV less than 8 cmH2O for at least 120 minutes, the nurses started to reduce End Expiratory Positive Pressure (PEEP) by 2cmH2O at a time to a maximum of 4cmH2O per day.
  When a patient was able to tolerate PSV less than 8 cmH2O with PEEP less than 6 cmH2O, the nurses started SBT trial: Continuos Positive Pressure Airways of 6cmH2O for at least 120 minutes and following discontinuation from ventilator.
  Groups: case

SUMMARY:
The purpose of this study is to evaluate the difference of the duration of weaning process from the ventilator between protocol-driven weaned patients and clinical judgment driven weaned patients.

DETAILED DESCRIPTION:
All patients with prolonged weaning and who required tracheostomy are enrolled in the study. These patients are randomized as "Case or Control" by a computer program.

Patients can start the weaning process when the acute phase of the respiratory failure has been resolved and pressure support ventilation was setted.

For all this patients are calculated modified-BWAP(BWAP-M) and TOBIN indexes. The "Case" patients started the weaning protocol process only if BWAP-M value is more than 15 or BWAP-M 10-15 with Tobin index < 100.

If not, the BWAP-M and Tobin will be calculated every day. The Control patients will start weaning by clinical judgement even if the BWAP-M value is less than 10.

For all patients are calculated: the duration of weaning process, the ICU length of stay and the duration of the mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. all patients that are clinically identified as prolonged to wean (failed 3 spontaneous breathing trials or 7 days or more of mechanical ventilation after the initial unsuccessful trial) and tracheostomized in ICU
2. improvement or resolution of the underlying causes of acute respiratory failure ratio between pressure partial artery of oxygen and fraction inspired oxygen (PaO2/FiO2) >200 with fraction inspired oxygen (FiO2)< 0,45.
3. pressure supported ventilation at the time of enrollment.

Exclusion Criteria:

1. patients assessed as easy weaning and not tracheostomized;
2. patients already tracheostomized on admission to ICU.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: difficult to wean patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
duration of weaning | within the first 15 days (plus or minus 5 days) after start of weaning

SECONDARY OUTCOMES:
duration of mechanical ventilation | within the first 12 days (plus or minus 10 days) after start of mechanical ventilation

OTHER OUTCOMES:
ICU length of stay | within the first 26 days (plus or minus 22 days) after ICU recovery
success of weaning | spontaneous breathing for 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Elena Peli, Principal Investigator
Locations (1):
- Institute of Anesthesiology and Intensive Care of the University of Brescia, Spedali Civili, Italy,, Brescia, Brescia, Italy